CLINICAL TRIAL: NCT05309499
Title: An Open, Prospective, Randomized Study on the Efficacy of Iron Therapy Using Intravenous (IV) Iron Supplements Relative to Oral Iron Intake for Increasing Left Ventricular Systolic Function in Patients With Myocardial Infarction
Brief Title: An Open Study on the Efficacy of Iron Therapy Using iv Iron Relative to Oral Iron for Increasing LV Systolic Function
Acronym: OPERA-MI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kazan State Medical University (Other)
Responsible Party: Principal Investigator, Dilyara Khastieva, Assistant Professor, PhD student, Kazan State Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BC2
Record Dates: First submitted 2022-03-24; First posted 2022-04-04 (Actual); Results first posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Myocardial Infarction; Iron-deficiency
Keywords: Myocardial Infarction; Iron-deficiency; WMSI; ferric carboxymaltose; left ventricular systolic function
MeSH Terms: conditions — Myocardial Infarction; Anemia, Iron-Deficiency | interventions — ferric carboxymaltose; ferrous sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FCM group (Active Comparator): The ferric carboxymaltose doses were determined using the patient's screening visit body weight measurement and haemoglobin value. Patients receives all doses during hospitalization accordance with the drug local labels.
  Interventions: Drug: ferric carboxymaltose
- Ferrous sulphate group (Active Comparator): 100 mg of ferrous sulphate is administrated 2 times per day during hospitalization and continue within next 2 month.
  Interventions: Drug: ferrous sulphate
- Group with normal iron status (No Intervention): Patiants with normal iron status

INTERVENTIONS:
Drug: ferric carboxymaltose — ferric carboxymaltose is i.v. iron, 99 patiants will be randomised to this group
  Arms: FCM group
Drug: ferrous sulphate — ferrous sulphate is oral iron, 100 patiants will be randomised to this group
  Arms: Ferrous sulphate group

SUMMARY:
The OPERA-MI trial evaluates the effect of i.v. ferric carboxymaltose compared to the effect of oral iron, on left ventricular systolic function.

DETAILED DESCRIPTION:
For this study an open-label prospective randomized approach is used. During the study 360 patients with or without ID, who hospitalized for myocardial infarction were signed up. Patients were randomised (1:1) to either intravenous. FCM or oral ferrous sulphate and received the treatment during hospitalisation. Patients are closely followed for 1 year. The primary outcome is a decrease in the Wall Motion Score Index value in FCM group compered to ferrous sulphate group. The main secondary outcome includes the composite of cardio-vascular mortality, non-fatal stroke, non-fatal MI, recurrent heart failure hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years of age) able to provide informed consent. Hospitalized myocardial infarction patients (that diagnosed according to Fourth Universal Definition of myocardial infarction and myocardial injury, ESC 2018) with hypokinesia or akinesia in at least two connected left ventricular segments according to echocardiography results obtained within the first 24 hours after myocardial infarction occurs.
* Hemoglobin >9.0 g/dL and <15,0 g/dl and serum iron <12 µmol/l on screening visit.
* Serum ferritin <100 μg/L, or 100-299 μg/L when transferrin saturation <20%.

Exclusion Criteria:

* Known hypersensitivity reaction to any component of ferric carboxymaltose.
* History of acquired iron overload, or the recent receipt (within 3 months) of erythropoietin stimulating agent, i.v. iron therapy, or blood transfusion.
* Heart failure Killip class II-IV on screening visit.
* Current or planned mechanical circulatory support or heart transplantation.
* Hemodialysis or peritoneal dialysis (current or planned within the next 6 months).
* Documented liver disease, or active hepatitis (i.e. alanine transaminase or aspartate transaminase >3 times the upper limit of normal range).
* Current or recent (within 3 years) malignancy with exception of basal cell carcinoma or squamous cell carcinoma of the skin, or cervical intraepithelial neoplasia.
* Active gastrointestinal bleeding.
* Female participant of child-bearing potential who is pregnant, lactating, or not willing to use adequate contraceptive precautions during the study and for up to 5 days after the last scheduled dose of study medication.
* Inability to return for follow up visits within the necessary period of time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2021-12-05 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kazan State Medical Universety, Kazan', Tatarstan Republic, Russia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- FCM Group: The ferric carboxymaltose doses were determined using the patient's screening visit body weight measurement and haemoglobin value. Patients receives all doses during hospitalization accordance with the drug local labels.
  ferric carboxymaltose: ferric carboxymaltose is i.v. iron, 121 patiants will be randomised to this group
- Ferrous Sulphate Group: 100 mg of ferrous sulphate is administrated 2 times per day during hospitalization and continue within next 2 month.
  ferrous sulphate: ferrous sulphate is oral iron, 121patiants will be randomised to this group
Period: Overall Study
Arm/Group | FCM Group | Ferrous Sulphate Group | Group With Normal Iron Status
Started | 99 | 100 | 99
Completed | 99 | 100 | 99
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FCM Group | Ferrous Sulphate Group | Group With Normal Iron Status | Total
Number analyzed (Participants) | 99 | 100 | 99 | 298
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (10.2) | 64.3 (8.8) | 66.1 (10) | 65.7 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 40 | 24 | 113
  Male | 50 | 60 | 75 | 185
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 99 | 100 | 99 | 298
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Decrease in the Wall Motion Score Index
Description: Using a standard transthoracic echocardiography sequence, each myocardial segment is assigned a score from 1 to 3. we used the 16 segment model of myocardial segmentation
  Each segment is then scored, using the following criteria:
  normokinesia (1 point) normal wall thickening and endocardial excursion hypokinesia (2 points) reduced wall thickening, reduced endocardial excursion akinesia (3 points) The wall motion score index is then calculated by dividing the sum of the aforementioned segmental values by the number of myocardial segments (16). A WMSI of 1.0 (16/16) is considered normokinetic, and correlates with a CMRI calculated ejection fraction of 64%, whereas a WMSI of 3.0 correlates with an ejection fraction of 12% and is considered akinetic. There are no spetial units of measure for it.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | FCM group | Ferrous sulphate group | Group with normal iron status
Number analyzed (Participants) | 99 | 100 | 99
Participants | 53 | 58 | 46

2. Secondary Outcome: Composite Outcome
Description: composite of cardio-vascular (CV) mortality, non-fatal stroke, non-fatal MI, recurrent HF hospitalizations.
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | FCM Group | Ferrous Sulphate Group | Group With Normal Iron Status
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/100 | 0/99
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/100 | 0/99
Other Adverse Events (participants affected / at risk) | 0/99 | 0/100 | 0/99

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT05309499/Prot_SAP_000.pdf